CLINICAL TRIAL: NCT05275790
Title: Electrical Vestibular Nerve Stimulation (VeNS) Together With a Lifestyle Modification Program, Compared to a Sham Control With a Lifestyle Modification Program, as a Means of Reducing Excess Body Weight.
Brief Title: Efficacy of Electrical Vestibular Nerve Stimulation (VeNS) in the Management of Obesity: A Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neurovalens Ltd. (Industry)
Collaborators: RD Gardi Medical College (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IVSWL001
Record Dates: First submitted 2022-02-02; First posted 2022-03-11 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Bilateral electrical vestibular nerve stimulation will be administered using a battery-powered vestibular nerve stimulator (ML 1000). Participants will act as their own self-control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vestal active device (Experimental): 10 subjects to receive an active device plus a diet plan for 12 weeks.
  Interventions: Device: Vestal device; Behavioral: Lifestyle intervention

INTERVENTIONS:
Device: Vestal device — Battery powered non-invasive neurostimulation device
Behavioral: Lifestyle intervention — All subjects will be prescribed a diet plan and instructed to follow it for the duration of the 12-week study. The diet plan will be designed by the P.I. who is a qualified, obesity management coach.

SUMMARY:
The aim of this study is to observe the efficacy of electrical vestibular nerve stimulation in the management of obesity.

Allocation: Active device (participants act as their own self-control) Endpoint classification: Efficacy Study. The study provides further evidence for the efficacy of electrical vestibular nerve stimulation in the management of obesity.

ELIGIBILITY:
Inclusion Criteria:

* BMI 30 to 40 kg/m2
* Aged above 18 years

Exclusion Criteria:

* Current use of any medications or therapy including use of oral contraceptives
* Use of dietary supplements known to affect the BMI
* Ear problems (assessed during physical examination)
* Any severe complications
* Unwilling participants

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-10-17 (Actual); Study Completion 2022-10-17 (Actual)

PRIMARY OUTCOMES:
Lipid profile | 12 weeks
  Blood sample to calculate ratio of Total Cholesterol: HDL and LDL

SECONDARY OUTCOMES:
Liver function tests | 12 weeks
  Albumin test
Complete blood count | 12 weeks
  Complete blood count
Glycated hemoglobin | 12 weeks
  HbA1c as a percentage
Mean blood glucose | 12 weeks
  Fasting glucose in mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Dr Sai Sailesh Kumar Goothy, Principal Investigator — RD Gardi Medical College, Ujjain
Locations (1):
- RD Gardi Medical College, Ujjain, Madhya Pradesh, India